CLINICAL TRIAL: NCT04366219
Title: Impact of Confinement and Preventive Measures in Period of SARS-COV2 Infection on Clinical Features, Diagnostic and Therapeutic Management and Prognosis of Patients With Lung Cancer: an Ambispective Study Extended Over 2 Time Periods.
Brief Title: Impact of Confinement and Preventive Measures in Period of SARS-COV2 Infection on Clinical Features, Diagnostic and Therapeutic Management and Prognosis of Patients With Lung Cancer
Acronym: CBP-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: ONCO PAYS de la LOIRE (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S15/03
Record Dates: First submitted 2020-04-27; First posted 2020-04-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-03

CONDITIONS: COVID; SARS-CoV 2; Lung Cancer
Keywords: Diagnostic management; Therapeutic management
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2019: Data collection on patients with Lung cancer diagnosed between March 13, 2019 and August 28, 2019.
- 2020: Data collection on patients with Lung cancer diagnosed between March 13, 2020 and August 28, 2020.

SUMMARY:
The unexpected onset of SARS-COV2 infection modified our practices, especially in routine medicine. In order to reverse the epidemic curve of severe cases and slow the spread of the infection, confinement was generalized in France from March 13, 2020.These restrictive measures were imposed on anyone with symptoms compatible with the infection, with the exception of dyspnea and other criteria of severity. March 12, 2020 is the pivotal date when the management of COVID came to interfere with medical and healthcare organizations. From this date, it is likely that some imaging or endoscopic exams have been de-scheduled for symptoms that are sometimes wrongly judged to be non-urgent and have seen their numbers drop dramatically.Otherwise, concerning lung cancer, preventive measures have been extremely strengthened. For instance, it is recommended to delay surgeries for localized tumors, to relieve or remove some chemotherapy or to delete radiotherapy sessions deemed non-essential. However, symptoms that may initially be attributed to viral infection, such as cough, fever, fatigue, or chest pain may be clinical indicators of early-stage Lung cancer. In addition, lung cancer is likely to make the patient more susceptible to pneumopathy, due to a weakened of immune response to viruses and bacteria. Consequently, as necessary as the restriction measures are, a risk of slowing down in the management of the Lung cancer pathology exists.

The CBP-COVID Study intends to assess consequences of restrictive measures linked to the SARS-COV2 epidemic, by comparing clinical characteristics at diagnosis, treatment times and treatments, regarding to 2 distinct time periods identical to the calendar, but one in 2019, the other in 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly diagnosed with a lung cancer based on histological or cytological criteria.
* Patient followed by investigating site participating in the study.
* Patient informed verbally and by an information document specifying the interest of the study and having given his oral agreement for the participation for the prospective part of the study.

Exclusion Criteria:

* Patient investigated and / or monitored in a site not involved in the study.
* Patient with lung cancer of incidental finding during hospitalization for another reason.
* Patient with recurrence of a previoulsy known lung cancer.
* Patient included in a clinical research trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 2019: Patient diagnosed with lung cancer from March 13, 2019 until August 28, 2019 Group 2020: Patient diagnosed with lung cancer from March 13, 2020 until August 28, 2020
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical characteristics | At the end of the second period, i.e. on August 28, 2020
  Comparison Group 2019 versus Group 2019

SECONDARY OUTCOMES:
Comparison of diagnostic procedures | At the end of the second period, i.e. on August 28, 2020
  Comparison Group 2019 versus Group 2020
Comparison of treatments (according to stage of disease) | At the end of the second period, i.e. on August 28, 2020
  Comparison Group 2019 versus Group 2020
Comparison of patients management deadlines | At the end of the second period, i.e. on August 28, 2020
  Comparison Group 2019 versus Group 2020
Comparison of survival | After 2 years post diagnoses
  Comparison Group 2019 versus Group 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France